CLINICAL TRIAL: NCT05392283
Title: Vacuum Cupping for Chronic Neck and Back Pain - a Feasibility Study
Brief Title: Vacuum Cupping for Chronic Neck and Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: University of Jena (Other); Helheten Norway (Unknown); National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Responsible Party: Principal Investigator, Winfried Meißner, Principal investigator, Jena University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC2022-1.0
Record Dates: First submitted 2022-04-26; First posted 2022-05-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Neck Pain; Back Pain
Keywords: Vacuum cupping; Quantitative sensory testing
MeSH Terms: conditions — Chronic Pain; Neck Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vacuum cupping (Experimental)
  Interventions: Device: AERO vacuum cupping device

INTERVENTIONS:
Device: AERO vacuum cupping device — The treatment consists of 5 sessions (approx. 30 min) of vacuum massage. The vacuum pump provided by the device provides a type of vacuum massage, that can be adjusted according to applied suction and air flow. The resulting massage technique provides a type of soft tissue manipulation similar to the ancient traditional medicine technique of cupping. Nonetheless, this automated technique allows for more precise determination of the massage characteristics.

SUMMARY:
Small clinical pilot studies have shown that vacuum massage-related techniques such as traditional dry cupping can reduce musculoskeletal pain such as back and neck pain. At the same time, little is yet known about the potential mechanisms of action of these therapies. A vacuum pump induces a massaging effect of the skin including the deeper tissue layers. The resulting massage technique corresponds to a kind of tissue manipulation similar to dry cupping. In this procedure, suction force and air flow can be individually adjusted. This is an advantage that can be used for patients with varying degrees of sensitivity or who are preloaded by patients with varying degrees of sensitivity or a history of pain. The aim of this study was to test the feasibility of the study design.

ELIGIBILITY:
Inclusion Criteria:

* chronic neck or back pain
* mean pain intensity ≥ 40 mm VAS

Exclusion Criteria:

* neurological symptoms or neuropathic pain
* vertebral column surgery less than 12 months prior to the study
* TENS, acupuncture, osteopathy, or a chiropractic maneuvre or infiltration at the area within 4 weeks prior to the inclusion in the study
* congenital deformation of the spine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity (Numeric rating scale (NRS)) | measured at baseline (week 1) and weekly during treatment (week 2 to 5) and 1 month after last treatment
  NRS is a 11-point pain scale for self-reporting of pain ("0" meaning "no pain" and "10" meaning "worst pain")

SECONDARY OUTCOMES:
Quantitative sensory testing (QST) | measured at baseline (week 1) and weekly during treatment (week 2 to 5) and 1 month after last treatment
  QST is a diagnostic tool which allows measurement of pain sensitivity.
Neck Disability Index (NDI) | measured at baseline (week 1), at the end of treatment (week 5) and after 1 month after last treatmentekly during treatment (week 2 to 5) and 1 month after last treatment
  NDI is used to measure neck pain and to quantify disability for neck pain.
Oswestry Disability Index (ODI) | measured at baseline (week 1), at the end of treatment (week 5) and after 1 month after last treatment
  ODI is used to measure low back pain and to quantify disability for low back pain.
Pain diary | filled in from baseline (week 1) until last treatment (week 5)
  A pain diary helps to track pain in the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Jena University Hospital, Jena, Germany

IPD SHARING:
Plan to Share IPD: Undecided